CLINICAL TRIAL: NCT00110643
Title: CoolTouch Non-ablative Laser Therapy for Acne Vulgaris
Brief Title: Infrared Non-Cutting Laser Therapy for Acne
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey S. Orringer, Professor of Dermatology, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Derm 494
Record Dates: First submitted 2005-05-11; First posted 2005-05-12 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Acne Vulgaris
Keywords: Acne; laser
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CoolTouch II laser

SUMMARY:
The purpose of this research project is to study the effect of non-ablative (non-cutting) laser therapy, a technique that uses laser energy to try to improve the appearance of the skin. In this study, we are interested in learning how well such a laser works to improve the symptoms of acne. The laser used in this particular study will be the CoolTouch II® laser, manufactured by ICN Photonics, Inc., and has not been FDA-approved for the treatment of acne.

DETAILED DESCRIPTION:
The purpose of this research project is to study the effect of non-ablative (non-cutting) laser therapy, a technique that uses laser energy to try to improve the appearance of skin. This type of laser treatment creates changes in a layer of the skin called the dermis without causing an open wound in the skin. It is not yet clear how much improvement can be seen with these treatments or exactly how the skin's response causes these improvements. In this study, we are interested in learning how well such a laser works to improve the symptoms of acne. The laser used in this particular study will be the CoolTouch II® laser, manufactured by ICN Photonics, Inc., and has not been FDA-approved for the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years or older of either gender and of any racial/ethnic group.
* Subjects must have clinically evident acne vulgaris of the facial skin.
* Subjects must understand and sign the informed consent prior to participation.
* Subjects must be in generally good health.
* Subjects must be able and willing to comply with the requirements of the protocol.
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* Oral retinoid (Accutane) use within 1 year of entry into the study.
* Systemic acne therapies (oral antibiotics) within 4 weeks of entry into the study.
* Topical acne therapies (retinoids, antibiotics) within 2 weeks of entry into the study.
* Microdermabrasion or superficial chemical peels at the sites to be treated within 3 months of entry into the study.
* Subjects with a history of dermabrasion or laser resurfacing at the sites to be treated.
* Use of topical lipid absorbing substances (Clinac AC) within 2 weeks of entry into the study.
* Non-compliant subjects.
* Subjects with a significant medical history or concurrent illness/condition which the investigator(s) feel is not safe for study participation.
* Subjects using alcohol-based topical solutions or "exfolliating" agents within 2 weeks of entry into the study.
* Subjects with a history of very frequent herpes simplex infections of the face or with clinical evidence of active herpes simplex infections.
* History of keloid scar formation for subjects undergoing biopsies.
* Pregnant or nursing females.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2003-02; Study Completion 2005-12

PRIMARY OUTCOMES:
Number of subtypes of acne lesions including papules, pustules, cysts, open comedones, and closed comedones

SECONDARY OUTCOMES:
total area of sebum droplets measured using image analysis software

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Dermatology Department, Ann Arbor, Michigan, United States